CLINICAL TRIAL: NCT07291739
Title: A Clinical Evaluation of a Phakic Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Staar Surgical Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP18-01
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Myopia; Hyperopia; Astigmatism; Presbyopia
MeSH Terms: conditions — Myopia; Hyperopia; Astigmatism; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EDOF ICL (Other): Eyes treated EVO+ Visian and EVO+ Toric Implantable collamer lens with aspheric optic determined by their preoperative refraction
  Interventions: Device: Implantable Collamer Lens (ICL)

INTERVENTIONS:
Device: Implantable Collamer Lens (ICL) — EVO+ Visian Implantable Collamer Lens with Aspheric (EDOF) Optic models VTICM6/VTICH6 (TEDOF ICL) and VICM6/VICH6 (EDOF ICL)

SUMMARY:
The objective of this study is to evaluate the clinical performance of the STAAR EVO+ Visian™ Implantable Collamer® Lens with Aspheric (EDOF) Optic as refractive elements to correct or reduce myopia or hyperopia with presbyopia with or without astigmatism.

DETAILED DESCRIPTION:
This prospective, open-labeled, evaluation of clinical performance of the investigational EDOF and Toric EDOF (TEDOF) ICL will be conducted at a single site in the Philippines.

Up to 45-50 subjects (90 eyes) who meet all eligibility criteria will be assigned to one of the following treatment arms, as determined by their preoperative refraction and the Investigator's medical judgement:

* EDOF Toric ICL in both eyes,
* EDOF Toric ICL in one eye and EDOF spherical ICL in fellow eye,
* EDOF spherical ICL in both eyes (up to 20 subjects/40 eyes).

Postoperatively, subjects will undergo ophthalmic examination at regular intervals per the study visit schedule up to 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Require a spherical lens power from -18.00 Diopters to +3.00 Diopters in both eyes or (in case of EDOF Toric) additional cylindrical lens power between +1.0 to +3.0 Diopters of Cylinder.
* Stable refractive history (+/-0.50 Diopters) as determined by manifest spherical equivalent.
* Requires +1.00 Diopters to +2.50 Diopters reading add in both eyes.
* Minimum distance corrected near visual acuity of 20/40 or worse in both eyes.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* History of previous ocular surgery.
* Progressive sight threatening disease.
* Low/abnormal endothelial cell density.
* Monocular.
* Serious acute non-ophthalmic disease.
* Pregnant or nursing women, or those who plan to become pregnant over the course of the study.
* Other protocol-specified exclusion criteria may apply.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Change in visual acuity | 1 month, 3 months and 6 months postoperatively
  Change from baseline in uncorrected distance, intermediate and near visual acuity and distance corrected near visual acuity
Change in refractive cylinder | 1 month, 3 months and 6 months postoperatively
  Change from baseline in absolute magnitude of subjective refractive cylinder
Lens axis misalignment | 1 month, 3 months and 6 months postoperatively
  Proportion of lenses with axis misalignment compared to operative day
Rotational stability | 1 day, 1, week, 1 month, 3 months and 6 months postoperatively
  Rotational stability by assessment of IOL axis meridian compared to placement on day of surgery
Compromise in visual acuity | 6 months postoperatively
  Clinically significant compromise in visual acuity based on subject questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Eye Institute, Makati City, Philippines

IPD SHARING:
Plan to Share IPD: No